CLINICAL TRIAL: NCT07231796
Title: Naldemedine in Clinical Practice in Cancer Patients With Opioid Induced Constipation: Clinical Outcomes and Patient Experience
Acronym: NOCON
Status: Recruiting | Type: Observational
Sponsor: Professor Monique A. H. Steegers (Other)
Collaborators: Viatris Inc. (Industry)
Responsible Party: Sponsor-Investigator, Professor Monique A. H. Steegers, Prof dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: 2025.0837
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Cancer; Opioid Induced Constipation (OIC)
MeSH Terms: conditions — Neoplasms; Opioid-Induced Constipation | interventions — naldemedine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Naldemedine, an peripherally acting opioid antagonist — Participants will be treated with naldemedine 0.2 milligrams orally once daily as monotherapy for a duration of 14 consecutive days, following discontinuation of laxatives, as intervention for opioid-induced constipation (OIC).

SUMMARY:
This study looks at how well a medicine called naldemedine works for people with cancer who become constipated while taking opioids. Opioids are medications prescribed to treat persistent or severe pain. Opioids can slow down the bowel and make it hard to pass stool. About 6 out of 10 people who use opioids have constipation. Laxatives such as lactulose or macrogol are described to help with this problem. If laxatives do not work, doctors may use special medicines called opioid blockers that act only in the gut. These medicines help relieve constipation without reducing pain relief. Naldemedine is one of these opioid blockers. It became available in the Netherlands in 2024 but is not yet widely used. The goal of this study is to learn how well naldemedine works in everyday care and how people feel while using it. Researchers will collect information on both medical results and participants' experiences.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* A diagnosis of malignancy
* Daily use of opioids
* Use of laxatives
* Experiencing constipation, defined as a Bowel Function Index (BFI) score ≥30
* Able to complete a Dutch-language questionnaire
* Able to provide written informed consent

Exclusion Criteria:

* Use of other opioid antagonists in the last month
* Suspected (risk of) gastrointestinal perforation
* Participation in another study that may confound the results of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be adults with cancer who are treated with opioids for pain managment. They will be recruited from multiple hospitals in the Netherlands. All participants will already be using laxatives to manage constipation. People who take part must be able to read Dutch and give written consent. Participants will represent a real-world group of individuals using opioids for cancer-related pain in daily clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
The change in Bowel Function Index (BFI) score | From enrollement to one week after initiation of naldemedine treatment
  Bowel Function Index (BFI) is a brief, three-item questionnaire assessing opioid-induced constipation over the past 7 days. It measures ease of defecation, sensation of incomplete evacuation and personal judgment of constipation, each rated on a 0-100 numerical rating scale. Scores are averaged and recalculated to a 0-100 scale; a score ≥30 indicates clinically significant opioid-induced constipation.

SECONDARY OUTCOMES:
The change in Bowel Function Index (BFI) score | From enrollment to two weeks after initiation of naldemedine
A clinically meaningful improvement in constipation | From baseline to one week after treatment initiation and from baseline to two weeks after treatment initiation.
  The proportion of patients achieving a ≥12-point decline in the Bowel Function Index (BFI) score.
The prevalence of persistent constipation, defined as a BFI score ≥ 30 | From enrollment to two weeks of treatment
The change in Patient Assessment of Constipation, Quality of Life (PAC-QoL) scores | From enrollment to two weeks of treatment with naldemedine
  The Patient Assessment of Constipation - Quality of Life (PAC-QoL) questionnaire is a 28-item questionnaire measuring the impact of constipation on daily functioning and well-being. Responses are given on a 5-point Likert scale, with higher scores indicating greater burden.
Continuation of naldemedine | From enrollment to two weeks after initiation of naldemedine
Patient Satisfaction | From enrollment to two weeks of treatment with naldemedine
  Patient satisfaction is measured on an 11-point Likert scale (0 = "Not satisfied at all", 10 = "Very satisfied").
Patient likelihood to recommend the use of naldemedine to other patients | From enrollment to two weeks of treatment with naldemedine
  Net Promoter Score (NPS): Based on the question: "How likely are you to recommend naldemedine to another patient?" (0 = "Not likely at all", 10 = "Very likely"). NPS is calculated as the percentage of promoters (scores 9-10) minus detractors (scores 0-6), yielding a score between -100 and +100.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided